CLINICAL TRIAL: NCT01626352
Title: Phase II Study of Bendamustine and Ofatumumab in Elderly Patients With Newly Diagnosed Diffuse Large B-Cell Lymphoma Who Are Poor Candidates for R-CHOP Chemotherapy
Brief Title: Study of Bendamustine and Ofatumumab in Elderly Patients With Newly Diagnosed Diffuse Large B-Cell Lymphoma Who Are Poor Candidates for R-CHOP Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Novartis (Industry); GlaxoSmithKline (Industry); Cephalon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LYM 75
Record Dates: First submitted 2012-06-20; First posted 2012-06-22 (Estimated); Results first posted 2017-10-18 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-10

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: Diffuse Large B-Cell Lymphoma; Ofatumumab; Bendamustine
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Bendamustine Hydrochloride; ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bendamustine/Ofatumumab (Experimental): All patients in this study will receive ofatumumab and bendamustine as an IV infusion for 6 cycles (a cycle is defined as 21 days in length). Patients will receive as an IV infusion of bendamustine Days 1 and 2 of Cycles 1-6, ofatumumab Days 1 and 8 during Cycle 1 only and on Day 1 of Cycles 2-6.
  Interventions: Drug: Bendamustine; Drug: Ofatumumab

INTERVENTIONS:
Drug: Bendamustine — Patients will receive as an IV infusion bendamustine 90 mg/m^2 Days 1 and 2 of Cycles 1 through 6.
  Other Names: Treanda
Drug: Ofatumumab — Patients will receive as an IV infusion ofatumumab 1000-mg IV Days 1 and 8 during Cycle 1 only, and on Day 1 of Cycles 2 through 6

SUMMARY:
This is a single-arm, Phase II study designed to enroll and treat up to 64 patients. All patients in this study will receive ofatumumab and bendamustine as an IV infusion for 6 cycles (a cycle is defined as 21 days in length). Patients will receive as an IV infusion bendamustine Days 1 and 2 of Cycles 1 through 6 and ofatumumab Days 1 and 8 during Cycle 1 only and on Day 1 of Cycles 2 through 6.

DETAILED DESCRIPTION:
While R-CHOP has improved survival and is considered standard of care for patients with DLBCL, the toxicities associated with R-CHOP are substantial in the elderly population. This is one of several reasons the outcome of older patients is worse than the corresponding younger patients. Bendamustine is an alkylating agent which causes intra- and inter-strand cross-links between DNA bases. Ofatumumab is a fully human anti-CD 20 antibody well tolerated by elderly patients. Ofatumumab targets a novel epitope of the CD20 molecule on B cells and remains on the cell surface twice as long as rituximab. The combination of both agents allows for a potentially efficacious, less toxic regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed CD20-positive DLBCL.
2. Newly diagnosed, stage III-IV DLBCL considered poor candidates for R-CHOP.
3. Age >=70 years
4. At least one of the following criteria:

   * ECOG PS 2
   * Cardiac compromise precluding anthracycline therapy
   * Previous anthracycline therapy for other malignancy precluding further anthracycline therapy.
   * Severe coexisting medical problems
   * General frailty
5. ECOG 0-2
6. Measurable disease with at least one bidimensional lymph node or tumor mass >1.5 cm in the longest diameter that can be followed for response as a target lesion as measured by CT
7. Patients must be HBV sAg and HBV cAb negative within 6 weeks of screening.
8. Patient must understand and voluntarily sign the IRB-approved informed consent.
9. Life expectancy >= 3 months
10. Laboratory parameters:

    * Absolute neutrophil count >=1,000 cells/mm3
    * Platelet count >=75,000 cells/mm3
    * Hemoglobin >=8 g/dL
    * Creatinine <=2.0 mg/dL or Creatinine Clearance >= 40 mL/min (calculated or 24 hour urine sample)
    * AST/SGOT <=2.0 x ULN (<=5.0 x ULN if secondary to lymphoma)
    * ALT/SGPT <=2.0 x ULN (<=5.0 x ULN if secondary to lymphoma)
    * Bilirubin level of <2.0 mg/dL unless secondary to Gilbert's disease (or pattern consistent with Gilbert's)

Exclusion Criteria:

1. Patients with active/symptomatic central nervous system (CNS) involvement based on clinical evaluation by lumbar puncture, PET, CT or MRI.
2. Known sensitivity to bendamustine or any component of bendamustine.
3. Known anaphylaxis or sensitivity to ofatumumab.
4. Major surgery within 28 days of Cycle 1, Day 1. Patients undergoing minor surgery within 7 days of Cycle 1, Day 1. (no wait needed for port placement)
5. Prior chemotherapy, immunotherapy, or irradiation for lymphoma.
6. Prior use of investigational anti-cancer agents for lymphoma.
7. HIV-related lymphoma.
8. Known active HIV or HCV infection, or known seropositivity for HIV, or current or chronic HBV or HCV infection. HBV test required at screening or a negative result within 6 weeks of screening.
9. Concurrent active or history of other malignancies, except non-melanoma skin cancer or carcinoma in situ of cervix or breast. Patients with previous malignancies are eligible provided they have been treated with curative intent and disease free for >= 1 year.
10. Serious (grade 3-4), active, intercurrent infection requiring therapy, or deep seated or systemic mycotic infections.
11. Myocardial infarction within 6 months prior to registration or New York Hospital Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or significant conduction system abnormalities, in the judgment of the Investigator.
12. Concurrent uncontrolled serious medical or psychiatric conditions likely to interfere with participation in this clinical study, in the judgment of the Investigator
13. Patients who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment).
14. Treatment with any known non-marketed drug substance or experimental therapy within 5 terminal half lives or 4 weeks prior to enrollment, whichever is longer, or currently participating in any other interventional clinical study.
15. Significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease which in the opinion of the investigator may represent a risk for the patient.
16. Male patients unable or unwilling to use adequate contraception methods from study start to one year after the last dose of protocol therapy.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Flinn, MD, PhD, Study Chair — SCRI Development Innovations, LLC
Locations (11):
- United States (11):
  - Florida Cancer Specialists-South, Fort Myers, Florida
  - Woodlands Medical Specialists, Pensacola, Florida
  - Florida Cancer Specialists North, St. Petersburg, Florida
  - Space Coast Cancer Center, Titusville, Florida
  - Providence Medical Group, Terre Haute, Indiana
  - RHHP/Hope Cancer Center, Terre Haute, Indiana
  - Grand Rapids Oncology Program, Grand Rapids, Michigan
  - Cancer Centers of Southwest Oklahoma, Lawton, Oklahoma
  - Oklahoma University, Oklahoma City, Oklahoma
  - Tennessee Oncology-Chattanooga, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee

REFERENCES:
- [Background] Aapro MS, Cameron DA, Pettengell R, Bohlius J, Crawford J, Ellis M, Kearney N, Lyman GH, Tjan-Heijnen VC, Walewski J, Weber DC, Zielinski C; European Organisation for Research and Treatment of Cancer (EORTC) Granulocyte Colony-Stimulating Factor (G-CSF) Guidelines Working Party. EORTC guidelines for the use of granulocyte-colony stimulating factor to reduce the incidence of chemotherapy-induced febrile neutropenia in adult patients with lymphomas and solid tumours. Eur J Cancer. 2006 Oct;42(15):2433-53. doi: 10.1016/j.ejca.2006.05.002. Epub 2006 Jun 5. PMID 16750358
- [Background] Cheson BD, Pfistner B, Juweid ME, Gascoyne RD, Specht L, Horning SJ, Coiffier B, Fisher RI, Hagenbeek A, Zucca E, Rosen ST, Stroobants S, Lister TA, Hoppe RT, Dreyling M, Tobinai K, Vose JM, Connors JM, Federico M, Diehl V; International Harmonization Project on Lymphoma. Revised response criteria for malignant lymphoma. J Clin Oncol. 2007 Feb 10;25(5):579-86. doi: 10.1200/JCO.2006.09.2403. Epub 2007 Jan 22. PMID 17242396
- [Background] Ansell SM, Falkson G, van der Merwe R, Uys A. Chronological age is a multifactorial prognostic variable in patients with non-Hodgkin's lymphoma. Ann Oncol. 1992 Jan;3(1):45-50. doi: 10.1093/oxfordjournals.annonc.a058068. PMID 1606068
- [Background] Armitage JO, Potter JF. Aggressive chemotherapy for diffuse histiocytic lymphoma in the elderly: increased complications with advancing age. J Am Geriatr Soc. 1984 Apr;32(4):269-73. doi: 10.1111/j.1532-5415.1984.tb02020.x. PMID 6368652
- [Background] Balducci L, Repetto L. Increased risk of myelotoxicity in elderly patients with non-Hodgkin lymphoma. Cancer. 2004 Jan 1;100(1):6-11. doi: 10.1002/cncr.11861. No abstract available. PMID 14692018
- [Background] Chang JE, Seo S, Kim KM, Werndli JE, Bottner WA, Rodrigues GA, Sanchez FA, Saphner TJ, Longo WL, Kahl BS. Rituximab and CHOP chemotherapy plus GM-CSF for previously untreated diffuse large B-cell lymphoma in the elderly: a Wisconsin oncology network study. Clin Lymphoma Myeloma Leuk. 2010 Oct;10(5):379-84. doi: 10.3816/CLML.2010.n.071. PMID 21030351
- [Background] Chow KU, Sommerlad WD, Boehrer S, Schneider B, Seipelt G, Rummel MJ, Hoelzer D, Mitrou PS, Weidmann E. Anti-CD20 antibody (IDEC-C2B8, rituximab) enhances efficacy of cytotoxic drugs on neoplastic lymphocytes in vitro: role of cytokines, complement, and caspases. Haematologica. 2002 Jan;87(1):33-43. PMID 11801463
- [Background] Coiffier B, Lepage E, Briere J, Herbrecht R, Tilly H, Bouabdallah R, Morel P, Van Den Neste E, Salles G, Gaulard P, Reyes F, Lederlin P, Gisselbrecht C. CHOP chemotherapy plus rituximab compared with CHOP alone in elderly patients with diffuse large-B-cell lymphoma. N Engl J Med. 2002 Jan 24;346(4):235-42. doi: 10.1056/NEJMoa011795. PMID 11807147
- [Background] Coiffier B, Radford J, Bosly A, Martinelli G, Verhoef G, Barca G, Davies A, Decaudin D, Gallop-Evans E, Padmanabhan-Iyer S, Van Eygen K, Wu KL, Gupta IV, Lin TS, Goldstein N, Jewell RC, Winter P, Lisby S; 415 study investigators. A multicentre, phase II trial of ofatumumab monotherapy in relapsed/progressive diffuse large B-cell lymphoma. Br J Haematol. 2013 Nov;163(3):334-42. doi: 10.1111/bjh.12537. Epub 2013 Aug 23. PMID 24032456
- [Background] Dixon DO, Neilan B, Jones SE, Lipschitz DA, Miller TP, Grozea PN, Wilson HE. Effect of age on therapeutic outcome in advanced diffuse histiocytic lymphoma: the Southwest Oncology Group experience. J Clin Oncol. 1986 Mar;4(3):295-305. doi: 10.1200/JCO.1986.4.3.295. PMID 3512783
- [Background] Feugier P, Van Hoof A, Sebban C, Solal-Celigny P, Bouabdallah R, Ferme C, Christian B, Lepage E, Tilly H, Morschhauser F, Gaulard P, Salles G, Bosly A, Gisselbrecht C, Reyes F, Coiffier B. Long-term results of the R-CHOP study in the treatment of elderly patients with diffuse large B-cell lymphoma: a study by the Groupe d'Etude des Lymphomes de l'Adulte. J Clin Oncol. 2005 Jun 20;23(18):4117-26. doi: 10.1200/JCO.2005.09.131. Epub 2005 May 2. PMID 15867204
- [Background] Habermann TM, Weller EA, Morrison VA, Gascoyne RD, Cassileth PA, Cohn JB, Dakhil SR, Woda B, Fisher RI, Peterson BA, Horning SJ. Rituximab-CHOP versus CHOP alone or with maintenance rituximab in older patients with diffuse large B-cell lymphoma. J Clin Oncol. 2006 Jul 1;24(19):3121-7. doi: 10.1200/JCO.2005.05.1003. Epub 2006 Jun 5. PMID 16754935
- [Background] Hainsworth JD, Flinn IW, Spigel DR, Clark BL, Griner PL, Vazquez ER, Doss HH, Shipley D, Franco LA, Burris HA 3rd, Greco FA; Sarah Cannon Oncology Research Consortium. Brief-duration rituximab/chemotherapy followed by maintenance rituximab in patients with diffuse large B-cell lymphoma who are poor candidates for R-CHOP chemotherapy: a phase II trial of the Sarah Cannon Oncology Research Consortium. Clin Lymphoma Myeloma Leuk. 2010 Feb;10(1):44-50. doi: 10.3816/CLML.2010.n.004. PMID 20223728
- [Background] Leoni LM, Bailey B, Reifert J, Bendall HH, Zeller RW, Corbeil J, Elliott G, Niemeyer CC. Bendamustine (Treanda) displays a distinct pattern of cytotoxicity and unique mechanistic features compared with other alkylating agents. Clin Cancer Res. 2008 Jan 1;14(1):309-17. doi: 10.1158/1078-0432.CCR-07-1061. PMID 18172283
- [Background] International Non-Hodgkin's Lymphoma Prognostic Factors Project. A predictive model for aggressive non-Hodgkin's lymphoma. N Engl J Med. 1993 Sep 30;329(14):987-94. doi: 10.1056/NEJM199309303291402. PMID 8141877
- [Background] Lipschitz DA. Age-related declines in hematopoietic reserve capacity. Semin Oncol. 1995 Feb;22(1 Suppl 1):3-5. No abstract available. PMID 7863350
- [Background] Ozer H, Armitage JO, Bennett CL, Crawford J, Demetri GD, Pizzo PA, Schiffer CA, Smith TJ, Somlo G, Wade JC, Wade JL 3rd, Winn RJ, Wozniak AJ, Somerfield MR; American Society of Clinical Oncology. 2000 update of recommendations for the use of hematopoietic colony-stimulating factors: evidence-based, clinical practice guidelines. American Society of Clinical Oncology Growth Factors Expert Panel. J Clin Oncol. 2000 Oct 15;18(20):3558-85. doi: 10.1200/JCO.2000.18.20.3558. No abstract available. PMID 11032599
- [Background] Pfreundschuh M, Schubert J, Ziepert M, Schmits R, Mohren M, Lengfelder E, Reiser M, Nickenig C, Clemens M, Peter N, Bokemeyer C, Eimermacher H, Ho A, Hoffmann M, Mertelsmann R, Trumper L, Balleisen L, Liersch R, Metzner B, Hartmann F, Glass B, Poeschel V, Schmitz N, Ruebe C, Feller AC, Loeffler M; German High-Grade Non-Hodgkin Lymphoma Study Group (DSHNHL). Six versus eight cycles of bi-weekly CHOP-14 with or without rituximab in elderly patients with aggressive CD20+ B-cell lymphomas: a randomised controlled trial (RICOVER-60). Lancet Oncol. 2008 Feb;9(2):105-16. doi: 10.1016/S1470-2045(08)70002-0. Epub 2008 Jan 15. PMID 18226581
- [Background] Strumberg D, Harstrick A, Doll K, Hoffmann B, Seeber S. Bendamustine hydrochloride activity against doxorubicin-resistant human breast carcinoma cell lines. Anticancer Drugs. 1996 Jun;7(4):415-21. doi: 10.1097/00001813-199606000-00007. PMID 8826610
- [Background] van Spronsen DJ, Janssen-Heijnen ML, Breed WP, Coebergh JW. Prevalence of co-morbidity and its relationship to treatment among unselected patients with Hodgkin's disease and non-Hodgkin's lymphoma, 1993-1996. Ann Hematol. 1999 Jul;78(7):315-9. doi: 10.1007/s002770050521. PMID 10466443
- [Background] Weidmann E, Kim SZ, Rost A, Schuppert H, Seipelt G, Hoelzer D, Mitrou PS. Bendamustine is effective in relapsed or refractory aggressive non-Hodgkin's lymphoma. Ann Oncol. 2002 Aug;13(8):1285-9. doi: 10.1093/annonc/mdf189. PMID 12181253
- [Background] Weidmann E, Neumann A, Fauth F, Atmaca A, Al-Batran SE, Pauligk C, Jager E. Phase II study of bendamustine in combination with rituximab as first-line treatment in patients 80 years or older with aggressive B-cell lymphomas. Ann Oncol. 2011 Aug;22(8):1839-44. doi: 10.1093/annonc/mdq671. Epub 2011 Jan 21. PMID 21257672
- [Derived] Flinn IW, Erter J, Daniel DB, Mace JR, Berdeja JG. Phase II Study of Bendamustine and Ofatumumab in Elderly Patients with Newly Diagnosed Diffuse Large B-Cell Lymphoma Who Are Poor Candidates for R-CHOP Chemotherapy. Oncologist. 2019 Aug;24(8):1035-e623. doi: 10.1634/theoncologist.2019-0286. Epub 2019 May 9. PMID 31073022

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between October 2012 to July 2014, 22 subjects with newly diagnosed Diffuse Large B-Cell Lymphoma (DLBCL) were screened for enrollment in the study at 12 investigational sites in the U.S.. Of those, 21 were treated.
Groups:
- Bendamustine/Ofatumumab: All patients will receive ofatumumab and bendamustine as an intravenous (IV) infusion for 6 cycles (a cycle is defined as 21 days in length).
  Bendamustine: via IV infusion, 90 mg/m^2 Days 1 and 2 of Cycles 1 through 6 Ofatumumab: via IV infusion, 1000-mg Days 1 and 8 during Cycle 1 only, and on Day 1 of Cycles 2 through 6
Period: Overall Study
Arm/Group | Bendamustine/Ofatumumab
Started | 22
Completed | 12
Not Completed | 10
Not completed — Disease Progression | 3
Not completed — Intercurrent Illness | 2
Not completed — Death | 2
Not completed — Withdrawal by Subject | 1
Not completed — Non-Compliance | 1
Not completed — Never Treated | 1

BASELINE CHARACTERISTICS:
Population: Includes all patients that received study drug.
Groups:
- Bendamustine/Ofatumumab: All patients in this study will receive ofatumumab and bendamustine as an IV infusion for 6 cycles (a cycle is defined as 21 days in length).
  Bendamustine: via IV infusion, 90 mg/m^2 Days 1 and 2 of Cycles 1 through 6 Ofatumumab: via IV infusion, 1000-mg IV Days 1 and 8 during Cycle 1 only and on Day 1 of Cycles 2 through 6
Arm/Group | Bendamustine/Ofatumumab
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 21
Age, Continuous [Median (Full Range); unit: years] | 83 [73 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With a Complete Response
Description: Disease response assessments will be performed using the International Working Group (IMW)-revised response criteria for malignant lymphoma (Cheson 2007). Complete response requires a disappearance of all evidence of disease.
Time Frame: 18 months
Population: All patients treated with study drugs and having a post baseline response assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Bendamustine/Ofatumumab
Number analyzed (Participants) | 21
Participants | 7

2. Secondary Outcome: Duration of Response
Description: Defined as the time from date of first documented confirmed response to date of disease progression or relapse from complete response as defined by the International Working Group (IMW)-revised response criteria for malignant lymphoma (Cheson 2007). This criteria categorizes the response of a patient's tumor to treatment as Complete Response (CR): the disappearance of all disease evidence; Partial Response (PR): regression of measurable disease and no new sites; Stable Disease (SD): less than a PR but not progressive disease (PD); Relapsed Disease or PD: Any new lesion or increase by ≥ 50% of previously involved sites from nadir. Patients who are alive and free from disease progression will be censored at the date of last tumor assessment. Patients who begin further anticancer therapy prior to disease progression will be censored at the date of last tumor assessment prior to the start date of the anticancer therapy.
Time Frame: After cycles 3 and 6 of each 21-day cycle and every 3 months thereafter until disease progression or relapse from complete response for up to 38 months
Population: All patients treated with study drugs and having a post baseline response assessment of a complete or partial response.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Bendamustine/Ofatumumab
Number analyzed (Participants) | 19
months | 5.6 [2.9 to 9.8]

3. Secondary Outcome: Time to Progression (TTP)
Description: Defined as the time from date of first treatment to the date of first documented disease progression or relapse from complete response as defined by the International Working Group (IMW)-revised response criteria for malignant lymphoma (Cheson 2007). This criteria categorizes the response of a patient's tumor to treatment as Complete Response (CR): the disappearance of all disease evidence; Partial Response (PR): regression of measurable disease and no new sites; Stable Disease (SD): less than a PR but not progressive disease (PD); Relapsed Disease or PD: Any new lesion or increase by ≥ 50% of previously involved sites from nadir.
Time Frame: After cycles 3 and 6 of each 21-day cycle, and every 3 months thereafter until progression or relapse from complete response for up to 40 months
Population: All enrolled patients who have received study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bendamustine/Ofatumumab
Number analyzed (Participants) | 21
months | 10.5 [4.5 to NA] — Not reached at this time

4. Secondary Outcome: Overall Survival (OS)
Description: Defined as the time from Day 1 of study drug administration to date of death from any cause.
Time Frame: every 3 cycles during treatment and every 3 months thereafter until progression or death from any cause, projected 18 months
Population: All enrolled patients who have received study treatment.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Bendamustine/Ofatumumab
Number analyzed (Participants) | 21
months | 12.0 [5.9 to 30.8]

5. Secondary Outcome: Overall Response (OR)
Description: Overall response is the number of patients with observed complete or partial response (CR or PR) as assessed using the International Working Group (IMW) revised response criteria for malignant lymphoma (Cheson 2007). Complete response requires disappearance of all evidence of disease. Partial response requires regression of measurable disease and no new sites.
Time Frame: after cycles 3 and 6 of each 21-day cycle, and every 3 months thereafter, projected 18 months
Population: All patients treated with study drugs and having a post baseline response assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Bendamustine/Ofatumumab
Number analyzed (Participants) | 21
Participants | 19

6. Secondary Outcome: Number of Patients With Treatment-Related Adverse Events (AEs) as a Measure of Safety
Description: A treatment-related adverse event was any untoward medical occurrence in a participant which was considered to have a relationship with the study drug (suspected to be possibly or probably related to the study drug per the Investigator's assessment). Adverse events were evaluated using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0.
Time Frame: after cycles 3 and 6 of each 21-day cycle, and up to 30 days after last dose, projected 24 weeks
Population: All enrolled patients who received the study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Bendamustine/Ofatumumab: All patients in this study will receive ofatumumab and bendamustine as an IV infusion for 6 cycles (a cycle is defined as 21 days in length). Patients will receive as an IV infusion of bendamustine Days 1 and 2 of Cycles 1-6, ofatumumab Days 1 and 8 during Cycle 1 only and on Day 1 of Cycles 2-6 (see Figure 1).
  Bendamustine: Patients will receive as an IV infusion bendamustine 90 mg/m^2 Days 1 and 2 of Cycles 1 through 6 and ofatumumab 1000-mg IV Days 1 and 8 during Cycle 1 only and on Day 1 of Cycles 2 through 6(a cycle is defined as 21 days in length).
  Ofatumumab: Patients will receive as an IV infusion bendamustine 90 mg/m^2 Days 1 and 2 of Cycles 1 through 6 and ofatumumab 1000-mg IV Days 1 and 8 during Cycle 1 only and on Day 1 of Cycles 2 through 6(a cycle is defined as 21 days in length).
Arm/Group | Bendamustine/Ofatumumab
Number analyzed (Participants) | 21
Participants | 16

7. Secondary Outcome: Progression-free Survival
Description: Defined as the time from first treatment until objective tumor progression, relapse from complete response, or death from any cause. Tumor response is defined by the International Working Group (IMW)-revised response criteria for malignant lymphoma (Cheson 2007). This criteria categorizes the response of a patient's tumor to treatment as Complete Response (CR): the disappearance of all disease evidence; Partial Response (PR): regression of measurable disease and no new sites; Stable Disease (SD): less than a PR but not progressive disease (PD); Relapsed Disease or PD: Any new lesion or increase by ≥ 50% of previously involved sites from nadir. Patients who are alive and free from disease progression will be censored at the date of last tumor assessment.
Time Frame: as for outcome 3
Population: All enrolled patients who have received study treatment.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Bendamustine/Ofatumumab
Number analyzed (Participants) | 21
months | 8.6 [4.6 to 10.6]

ADVERSE EVENTS:
Time Frame: Collected once per week during cycle 1 and then collected once per month until 30 days after last treatment.
Description: All patients who received at least one dose of protocol treatment are included in the safety analysis.
Arm/Group | Bendamustine/Ofatumumab
All-Cause Mortality (participants affected / at risk) | 14/21
Serious Adverse Events (participants affected / at risk) | 9/21
Other Adverse Events (participants affected / at risk) | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bendamustine/Ofatumumab (N=21)
Pulmonary Embolism (Vascular disorders) | 1
Deep Vein Thrombosis (Vascular disorders) | 1
Pneumonia (Infections and infestations) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal infection (Infections and infestations) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Cystitis (Infections and infestations) | 1
Death (General disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fatigue (General disorders) | 1
Gastrointestinal necrosis (Gastrointestinal disorders) | 1
Haemoglobin decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Syncope (Nervous system disorders) | 1
Urinary tract infection (Infections and infestations) | 1
White blood cell count decreased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bendamustine/Ofatumumab (N=21)
Fatigue (General disorders) | 10
Nausea (Gastrointestinal disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 5
Anaemia (Blood and lymphatic system disorders) | 4
Constipation (Gastrointestinal disorders) | 4
Decreased Appetite (Metabolism and nutrition disorders) | 4
Infusion Related Reaction (General disorders) | 4
Weight Decreased (Investigations) | 4
Oedema Peripheral (General disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Asthenia (General disorders) | 2
Chest Pain (Cardiac disorders) | 2
Headache (Nervous system disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypotension (Vascular disorders) | 2
Insomnia (Psychiatric disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 2
Neutrophil Count Decreased (Investigations) | 2
Platelet Count Decreased (Investigations) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.